CLINICAL TRIAL: NCT00214019
Title: The Effect of Salmeterol on Eosinophil (EOS) Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-2003-0469
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Diskus (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo
- Salmeterol Diskus 50 mcg twice per day (Experimental): Salmeterol Diskus 50 mcg twice per day
  Interventions: Drug: salmeterol
- Placebo diskus, fluticasone (Experimental): placebo diskus, fluticasone MDI 88 mcg twice per day
  Interventions: Drug: Fluticasone
- Salmeterol, Fluticasone (Experimental): Salmeterol diskus 50 mcg BID, fluticasone MDI 88 mcg twice per day
  Interventions: Drug: salmeterol; Drug: Fluticasone

INTERVENTIONS:
Drug: salmeterol — salmeterol diskus 50 mcg twice per day
  Other Names: Seravent; Advair
  Arms: Salmeterol Diskus 50 mcg twice per day; Salmeterol, Fluticasone
Drug: Fluticasone — placebo diskus, fluticasone MDI 88 mcg twice per day
  Other Names: flovent; advair
  Arms: Placebo diskus, fluticasone; Salmeterol, Fluticasone
Drug: Placebo — placebo diskus
  Other Names: no drug; comparator treatment
  Arms: Placebo Diskus

SUMMARY:
This study is designed to test the hypothesis that salmeterol use, and not fluticasone use or the combination treatment with fluticasone and salmeterol, is associated with a greater number of sputum eosinophils following antigen challenge and, under these circumstances, the migrating peripheral blood eosinophils are less adherent.

DETAILED DESCRIPTION:
An antigen challenge is when a participant inhales either cat, ragweed, or dust dander in increasing concentrations until their lung function drops 15 or 20 percent.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* history of asthma symptoms for the previous 6 months
* Forced Expiratory Value (FEV1) >75% of predicted
* positive prick skin test to cat, house dust mite or ragweed

Exclusion Criteria:

* history of life threatening asthma or anaphylaxis
* current smoker
* pregnant or breast-feeding
* evidence of an upper respiratory infection within 4 weeks of screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at UW Hospital and Clinics, Madison, WI from November 2003 to January 2008.
Pre-assignment Details: 6 participants completed all four arms of the study. 36 participants were recruited; 17 screen failed prior to randomization, 11 were lost to follow up prior to randomization, and 2 withdrew consent prior to randomization.
Groups:
- All Study Participants: All participants completed all 4 arms of the study. 28 days per arm.
Period: Overall Study
Arm/Group | All Study Participants
Started | 36
Placebo/Placebo Arm | 6
Placebo/Salmeterol Arm | 6
Fluticasone/Placebo Arm | 6
Fluticason/Salmeterol Arm | 6
Completed | 6
Not Completed | 30
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failed prior to randomization | 17

BASELINE CHARACTERISTICS:
Population: This is a randomized/double-blinded/placebo-controlled/four-phase/crossover trial in subjects with a history of mild allergic asthma. Treatment arms included placebo, fluticasone 44 µg twice daily, salmeterol 50 µµg twice daily and combined FT and SA treatment, all given by inhalers. The order of these treatments was randomized for each subject.
Groups:
- 4 Way Cross Over: Participants completed all 4 arms:
  Placebo, Salmeterol diskus 40 mcg twice per day, Placebo then fluticasone, Salmeterol then Fluticasone,
Arm/Group | 4 Way Cross Over
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Sputum Eosinophils (EOS) 24 Hours Post Antigen Challenge
Description: Sputum samples were collected from the participants. Cell counts were made from these samples after treatment with 0.1% dithiothreitol. Percentage of eosinophils were reported. Time frame measurement was 24 hours after the subject had an antigen challenge.
Time Frame: Eosinophils are measured 24 hours after the subject has an antigen challenge
Population: Participants for analysis included any subject that completed that specific treatment phase, even if they did not complete other treatment phases.
Measure: Mean (Standard Deviation); unit: Eosinophil percentage
Groups:
- Placebo/Placebo: Participants on Placebo/Placebo arm
- Placebo/Salmeterol: Participants on Placebo/Salmeterol arm
- Placebo/fFuticasone: Participants on Placebo/Fluticasone arm
- Salmeterol/Fluticasone: Participants on Salmeterol/Fluticasone
Arm/Group | Placebo/Placebo | Placebo/Salmeterol | Placebo/fFuticasone | Salmeterol/Fluticasone
Number analyzed (Participants) | 6 | 6 | 6 | 6
Eosinophil percentage | 3.5 (3.4) | 2.4 (3.4) | 0.54 (0.39) | 2.4 (2.6)

ADVERSE EVENTS:
Time Frame: 2.5 years
Description: Subject interview at visit
Groups:
- 4 Way Cross Over: Participants completed all 4 treatments:
  Placebo Salmeterol diskus 50 mcg twice per day Placebo then Fluticasone Salmeterol then Fluticasone
Arm/Group | 4 Way Cross Over
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 Way Cross Over (N=6)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ARM: Fluticasone/Placebo
Increased asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ARM: Placebo/Salmeterol
Back Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) — ARM: Fluticasone/Salmeterol
Scratchy throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ARM: Fluticasone/Placebo
Fainted (Vascular disorders) | 1 (1) — ARM: Fluticasone/Placebo

LIMITATIONS AND CAVEATS:
36 subjects were screened, identifying subjects with both a peripheral eosinophil count >0.200x106 cells/ml and a LPR >15% was more difficult than expected. Of the subjects screened, only 12 met criteria and 6 subjects completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No